CLINICAL TRIAL: NCT01877837
Title: Reduced Intensity Matched Sibling Bone Marrow Transplantation for Sickle Cell Anemia in Patients 2-30 Years Old
Brief Title: Stem Cell Transplantation for Sickle Cell Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001894
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Sickle Cell Disease
Keywords: Stem cell transplant; Sickle cell; Stem cell transplantation; Related; Unrelated
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; fludarabine; fludarabine phosphate; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Related donor (Experimental): Matched sibling donors (9-10/10 marrow/PBSC or 5-6/6 UCB (single) with a total TNC dose of greater than 5 x 107/kg recipient weight), age 2-30 years after conditioning regimen Alemtuzumab , Fludarabine, and Melphalan.
  1) Patients will receive a conditioning regimen composed of Alemtuzumab, Fludarabine, and Melphalan as detailed in the table below.
  Day Treatment
  * -22 Alemtuzumab 3mg IV (test dose)
  * -21 Alemtuzumab 10mg IV
  * -20 Alemtuzumab 15mg IV
  * -19 Alemtuzumab 20mg IV
  * -8 Fludarabine 30mg/m2 IV
  * -7 Fludarabine 30mg/m2 IV
  * -6 Fludarabine 30mg/m2 IV
  * -5 Fludarabine 30mg/m2 IV
  * -4 Fludarabine 30mg/m2 IV
  * -3 Melphalan 140mg/m2 IV
  * -2 Rest Day
  * -1 Rest Day
  * 0 Stem Cell Infusion
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Melphalan; Procedure: Stem Cells

INTERVENTIONS:
Drug: Alemtuzumab — Adjusted Ideal Body Weight Formula: AIBW = IBW + [(0.4) x (ABW - IBW)]
  b) Medications
  i.) Alemtuzumab I. Hb S% must be < or = 45% within 7 days prior to initiation of Alemtuzumab II. Iron chelation and hydroxyurea must be discontinued >48 hours before initiating therapy III. Alemtuzumab will be diluted in 100mL of 0.9% NS and infused at a rate as below
  Other Names: Alemtuzumab (Campath)
Drug: Fludarabine — I. Fludarabine should be diluted in 100 ml 0.9%NS and given over 30 minutes. II. A daily dose of an antiemetic should be given 30 minutes prior to administration of the Fludarabine
  Other Names: Fludarabine (Fludara)
Drug: Melphalan — I. Melphalan should be diluted in 0.9%NS to a concentration of 0.1 -0.45 mg/mL and given over 45 minutes. *Entire dose must be infused within 60 minutes of reconstitution in Pharmacy.
  II. A daily dose of an antiemetic should be given 30 minutes prior to administration of the Melphalan III. Patients should be encouraged to suck on a popsicle or something similar during the Melphalan infusion.
  Other Names: Melphalan (Alkeran)
Procedure: Stem Cells — Infusion of Hematopoietic Stem Cells

SUMMARY:
This protocol will be investigating the use of stem cell transplantation, in related donors, to cure sickle cell disease. Sickle cell disease is a recessive disorder caused by a point mutation that results in the substitution of valine for glutamic acid at the sixth position in the B-chain of hemoglobin. This leads to sickling of the red blood cells under many conditions, such as hypoxia, dehydration, and hyperthermia. The sickling leads to vaso-occlusion, which causes irreversible damage in almost all systems in the body, including the central nervous system (CNS), lungs, heart, bones, eyes, liver, and kidneys.

DETAILED DESCRIPTION:
Primary objective:

1) To determine disease free survival (DFS) at two years after matched sibling transplant using bone marrow (BM) after a conditioning regimen consisting of distal timed Alemtuzumab, Fludarabine, and Melphalan for patients 2-30 y/o

Secondary objectives:

1. Overall survival
2. Rate of neutrophil and platelet engraftment for BM
3. Incidence of graft failure
4. Incidence of grade II-IV and grade III-IV acute graft vs host disease (GVHD)
5. Incidence of chronic GVHD
6. Incidence of other transplant complications, such as veno-occlusive disease, central nervous system (CNS) toxicity, and idiopathic pneumonia syndrome (IPS)
7. Incidence of reactivation of CMV, EBV, adenovirus, BK/JC virus
8. Incidence of invasive fungal disease
9. Time to immune reconstitution via monitoring of lymphocyte subpopulations and immunoglobulin levels

ELIGIBILITY:
Inclusion Criteria:

* Patient Eligibility

  1) Matched sibling donors (9-10/10 marrow/PBSC or 5-6/6 UCB (single or double) with a total TNC dose of greater than 5 x 107/kg recipient weight)
  1. Age 2-30
  2. Hb SS, S-thal0, S-thal+, SC
  3. Evidence of ongoing hemolysis: Hb<10, retic >5%, LDH > 500, TB>2
  4. Karnofsky/Lansky score >50
  5. LVSF>26% or LVEF>40%
  6. DLCO >40% or O2 sat >85% for those patients that can't perform PFTs
  7. GFR >70 and serum creatinine < 1.5 * ULN for age
  8. ALT and AST < 5 x ULN, direct bilirubin <2 x ULN
  9. If the patient has been on chronic transfusion or has a ferritin >1000, liver biopsy should be done and show no evidence of bridging fibrosis or cirrhosis
* Exclusion criteria

  1. Evidence of uncontrolled bacterial, viral, or fungal infection within one month prior to initiation of the conditioning regimen
  2. Pregnant or breastfeeding
  3. HIV positive
  4. Written informed consent not obtained

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Krajewski, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Sickle Cell Anemia: Patients with sickle cell anemia, age 2-30, that received transplant after after conditioning regimen Alemtuzumab, Fludarabine, and Melphalan.
Period: Overall Study
Arm/Group | Patients With Sickle Cell Anemia
Started | 30
Completed | 25
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Population: Baseline information of patients that received transplant at the time of transplant.
Arm/Group | Patients With Sickle Cell Anemia
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.68 [2.25 to 25.42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity Information was not collected. Population: Race/Ethnicity Information was not collected.
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Graft Failure
Description: Primary endpoint:
  In each group, the Number of participants with Graft Failure at the 2 years endpoint will be estimated using the Kaplan Meier product limit estimator.
Time Frame: 2 years
Population: Patients that were followed at 2 years post transplant for graft failure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Sickle Cell Anemia
Number analyzed (Participants) | 23
Participants | 3

2. Secondary Outcome: Overall Survival
Description: Secondary endpoints:
  Overall survival: The distribution of time to death from any cause will be estimated by Kaplan- Meier product limit function and plotted. The overall survival will be measured from the time of transplant to any death and patients will be followed for 2 years.
Time Frame: 2 years
Population: Patients surviving at 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Sickle Cell Anemia
Number analyzed (Participants) | 25
Participants | 23

ADVERSE EVENTS:
Time Frame: 2 year post transplant
Description: Adverse events grade 3 and above (including deaths) were considered as serious adverse events and are reported
Arm/Group | Patients With Sickle Cell Anemia
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 13/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Sickle Cell Anemia (N=25)
Infection (grade 3 and above) (Infections and infestations) | 9 (9)
Renal insufficiency (Renal and urinary disorders) | 2 (2)
SupraVentricular Tachycardia (Cardiac disorders) | 1 (1)
Alerted mental status (Nervous system disorders) | 1 (1)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT01877837/Prot_SAP_000.pdf